CLINICAL TRIAL: NCT03336567
Title: Understanding Patients and Prescriber Perceptions of Cell and Gene Therapy (CGT) in Oncology
Brief Title: Perceptions of Cell and Gene Therapies (CGT) for the Treatment of Cancer
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 207202
Record Dates: First submitted 2017-11-05; First posted 2017-11-08 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Neoplasms
Keywords: telephonic interview; TCR Therapy; cross-sectional; CGT; qualitative
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Subjects with hematological malignancies: It will include subjects with Refractory Diffuse Large B-cell Lymphoma and Multiple Myeloma, Relapsed or Refractory Acute Lymphoblastic Leukemia (ALL) and/or who participated in a CAR-T clinical trial or autologous treatment. Subjects will undergo a telephonic interview for up to 90 minutes.
  Interventions: Other: Telephonic interview
- Subjects with NSCLC or soft-tissue sarcoma: It will Include subjects with NSCLC on second or later-line therapy or soft-tissue sarcoma on second or later line therapy. Subjects will undergo a telephonic interview for up to 90 minutes.
  Interventions: Other: Telephonic interview
- Oncologists from academic centers with CGT experience: It will include oncologists using TCR therapies, CAR-T or participating in CAR-T or TCR therapy clinical trials. Oncologists will undergo a telephonic interview for up to 60 minutes.
  Interventions: Other: Telephonic interview
- Oncologists from community clinics: It will include oncologists from community clinics who evaluate, prescribe, treat, and actively interact with subjects with NSCLC or soft tissue sarcoma, who have used immuno-oncology (IO) therapies. Oncologists will undergo a telephonic interview for up to 60 minutes.
  Interventions: Other: Telephonic interview

INTERVENTIONS:
Other: Telephonic interview — Subjects with cancer and Oncologists will undergo a semi-structured one-to-one telephonic interview for up to 90 and 60 minutes respectively.

SUMMARY:
Gene and cell therapies have a real value potential (example: potential long-term effect, curative potential, and single administration) but also drawbacks (example: treatment perceived as complex and risky generating fear and anxiety in subjects and their family; high cost) that require significant educational efforts and planning for optimal market access. It is therefore important to understand subject and physician perceptions of T-Cell Receptor (TCR) therapies. The aim of this study is to collect qualitative data from a small but diverse sample of oncologists and subjects in the United States to gather qualitative evidence for a preliminary understanding about their perceptions of T-cell therapies in the treatment of cancer. This cross-sectional study will involve up to 20 adult subjects with cancer and up to 20 oncologists/hematologist-oncologists in the United States. Eligible subjects will be scheduled for a telephone interview lasting approximately 60-90 minutes. Eligible oncologists will be scheduled for a telephone interview lasting approximately 60 minutes.

Searching social media is another way of understanding the perceptions of prescribers and consumers of CGT, in addition to interviews being conducted under the original protocol. The results of a feasibility assessment suggested that it would be helpful to explore social media to add to the findings from the interviews. This social media study(SMS) is being conducted as a pilot study to hone methods for future explorations of social media. The pilot study will investigate and describe initial themes emerging from existing discussions related to CGT. Findings from this work will help GlaxoSmithKline to plan future work in the social media landscape.

ELIGIBILITY:
Inclusion Criteria:

For cancer subjects:

* Adults 18 years of age and older of any, sex, racial/ethnic group, or economic status
* With a self-reported diagnosis of non-small-cell lung carcinoma (NSCLC), soft tissue sarcomas, or hematological malignancies
* Willing and able to participate in a telephone interview
* Willing to be audio-recorded during the interview session

For Oncologists:

* Education credentials equivalent to Doctor of Medicine (MD)
* Oncologist/hematologist-oncologist with at least five years of experience in oncology
* Able to fluently read, speak, and understand English to participate in an interview and/or complete all assessments
* Willing and able to participate in a telephone interview
* Willing to be audio-recorded during the interview session

Exclusion Criteria:

For cancer subjects:

* Diagnosed with cancer less than a year ago or those on first line of treatment at the time of the interview
* Unable to provide information on their line of treatment
* Significant speech impairment, cognitive impairment, hearing difficulty, visual impairment, or severe psychopathology (according to the opinion of the screener)
* Any clinically-relevant medical condition including, but not limited to, severe co-morbid condition, severe mental illness, substance abuse, cognitive, or other impairment (e.g., visual) which, in the opinion of the investigator, would interfere with participating in an interview and/or completing the study procedures.

For Oncologists:

* Currently unable to practice medicine and/or treat subjects, for reasons including (but not limited to): expired medical license, revoked medical license, or part of the Food and Drug Administration (FDA) debarment list.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A small but diverse convenience sample of up to 20 adult cancer subjects and 20 oncologists/hematologist-oncologists in the United States will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with feedback as having benefit of CGT during interview | Up to 90 minutes
  Telephonic interview will be conducted to assess preliminary understanding about subjects perceptions of CGT, especially TCR and CAR T-Cell therapies in the treatment of cancer.
Number of subjects with feedback as having concerns of CGT during interview | Up to 90 minutes
  Telephonic interview will be conducted to assess preliminary understanding about subjects perceptions of CGT, especially TCR and CAR T-Cell therapies in the treatment of cancer.
Number of subjects with feedback as having fear of CGT during interview | Up to 90 minutes
  Telephonic interview will be conducted to assess preliminary understanding about subjects perceptions of CGT, especially TCR and CAR T-Cell therapies in the treatment of cancer.
Number of subjects with willingness to be treated with CGTs | Up to 90 minutes
  Telephonic interview will be conducted to assess preliminary understanding about subjects perceptions of CGT, especially TCR and CAR T-Cell therapies in the treatment of cancer.
Number of physicians who would initiate potential referrals to utilize CGT therapies | Up to 60 minutes
  Telephonic interview will be conducted to assess preliminary understanding about physicians perceptions of CGT, especially TCR and CAR T-Cell therapies in the treatment of cancer.
Number of physicians with decisions to use CGT in subjects with cancer | Up to 60 minutes
  Telephonic interview will be conducted to assess preliminary understanding about physicians perceptions of CGT, especially TCR and CAR T-Cell therapies in the treatment of cancer.
Number of physicians with concerns to use CGT in subjects with cancer | Up to 60 minutes
  Telephonic interview will be conducted to assess preliminary understanding about physicians perceptions of CGT, especially TCR and CAR T-Cell therapies in the treatment of cancer.
Number of physicians with feedback as CGT sound better than other types of cancer treatments | Up to 60 minutes
  Telephonic interview will be conducted to assess preliminary understanding about physicians perceptions of CGT, especially TCR and CAR T-Cell therapies in the treatment of cancer.
Number of physicians with feedback as CGT sound more concerning than other types of cancer treatments | Up to 60 minutes
  Telephonic interview will be conducted to assess preliminary understanding about physicians perceptions of CGT, especially TCR and CAR T-Cell therapies in the treatment of cancer.
Number of physicians with feedback of recommending CGT in the future | Up to 60 minutes
  Telephonic interview will be conducted to assess preliminary understanding about physicians perceptions of CGT, especially TCR and CAR T-Cell therapies in the treatment of cancer.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Collegeville, Pennsylvania, United States